CLINICAL TRIAL: NCT01782521
Title: Is a Primer Needed for Orthodontic Bonding? A Multi-centre RCT
Brief Title: Is a Primer Needed for Orthodontic Bonding? A Multi-centre Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bradford Teaching Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Madeleine Storey, Speciality Registrar in Orthodontics, Bradford Teaching Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: primerstudy01
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Bracket Failure Rate; Bonding Time Per Bracket; Adhesive Remnant Index for Type of Bond Failure; Length of Treatment; Peer Assessment Rating
Keywords: Bracket failure rate; Orthodontic bonding; Primer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primer (No Intervention): Metal brackets bonded with primer
- No primer (Experimental): Metal brackets bonded without primer
  Interventions: Procedure: No primer

INTERVENTIONS:
Procedure: No primer — Primer not used when bonding orthodontic brackets
  Arms: No primer

SUMMARY:
Orthodontic treatment is carried out by placing fixed attachments(brackets)on teeth with wires which run through them and create tooth movement. These metal brackets are bonded (glued) onto the tooth surface by a three step process. Firstly, a mild acid is used to roughen the tooth surface, secondly a free flowing glue (composite primer) is used to fill in the roughened pores and thirdly, the bracket is glued on to the tooth surface with a 'composite' material which sets hard by exposure to a high intensity light.The success of this procedure is measured by bracket failure rates.

The literature review suggests that the scientific evidence is not clear to indicate whether the use of a primer is absolutely essential to achieve acceptable bracket success rates in a clinical environment.

The primary aim of the study is to find out if the rate of loss of orthodontic brackets is clinically acceptable when they are glued onto the tooth surface without the use of a primer as compared to brackets bonded with a primer over a 12 month study period. The investigators will also investigate the Bonding time,Type of bracket bond failure,length of treatment and Peer Assessment Rating scores (PAR)

This RCT will be undertaken on consented NHS patients in 3 hospitals in Yorkshire region by multiple operators

The results from this study will help improve our knowledge of the best approach to bonding metal brackets on teeth. If the bracket failure rate is similar in both groups, this would indicate that the use of a primer is not always necessary. For patients, this would mean lesser time required to place brackets at the start of orthodontic treatment. For clinicians and NHS purchasers the outcome will influence cost effectiveness (as the primer is the most expensive component in the bonding process) and provide a framework for future studies.

DETAILED DESCRIPTION:
AIMS OF THE TRIAL The primary aim of the trial is to find out if clinically acceptable bracket failure rates can be achieved when metal brackets (fixed brace attachments) are glued (bonded) to teeth without the use of a primer as compared to brackets glued with a conventional primer in adolescent and adult orthodontic patients over a 12 month study period.

The other objectives are to determine if the gluing time per bracket is different between the groups and the type of glue failure at bracket-tooth interface using Adhesive Remnant Index. Length of treatment time and Peer Assessment Rating scores will also be analysed.

HYPOTHESES The null hypothesis for the primary outcome is - "there is no difference in the bracket failure rates when metal brackets are bonded with primer as compared to those which are bonded without a primer".

The null hypotheses for the secondary outcomes are - "there is no difference in the bonding time per bracket and the type of bond failure using Adhesive Remnant Index between the control and experimental group in this study.

METHOD OF INVESTIGATION

1. Sample population All patients referred to the Leeds Dental Institute/Seacroft hospital/ St.Luke's hospital, Bradford who qualify for orthodontic treatment.
2. Setting Patients treated in a dental teaching hospital and district NHS hospital setting
3. Operator characteristics All patients will be treated from the start until the end of the study period by 6 operators of various experience (NHS specialist registrar at two sites - Leeds Dental Institute and St.Luke's Hospital, orthodontic therapists (SLH) and consultant orthodontists (SLH/LDI and Seacroft hospitals)
4. Study design A multicentre single-blinded randomised controlled clinical trial in a NHS hospital setting. Individual patients will be allocated randomly to either the test or control group.
5. Intervention Test group - Metal brackets will be bonded without a primer Control group - Metal brackets will be bonded with primer
6. Methods to minimise bias - Randomisation and Blinding All consecutive patients who need fixed appliance treatment will be taken off the waiting list and no attempt will be made to match them for age, sex or malocclusion to ensure a representative sample, except for the exclusion criteria. After informed consent is obtained, they will be randomly allocated to either the control (with primer) or experimental (without primer) group. This will be done by preparing opaque numbered sealed envelopes in blocks of 10 in advance by the supervisor (NH) using random number tables. The supervisor will enroll the participants and assign them to their group using the sealed envelopes which blinds the two operators and participants to the assignment before enrollment. Once the envelopes are opened the blinding of the operators will be lost. The operators cannot be blinded in this trial as the intervention administered to the test group cannot be blinded. Treatment will be started on all patients within 3 months of the enrollment.
7. Agreed start and end points Upper and lower teeth will be bonded when appropriate. If upper and lower teeth are bonded at separate visits, then the specific dates will be considered as the start point. The follow up period will be for 12 months and the incidence of first bracket loss will be recorded (i.e. event). Any subsequent bracket loss will also be recorded. For patients who have no failures the bracket survival time will be followed up until the end of fixed appliance treatment by the original or subsequent operator (i.e. anybody involved in the follow-up of these patients after the end of 12 month study period). In the event of repeated failures in the same patient or in the same area, the data will be recorded and statistical analysis for clustering will be appropriately selected.
8. Subject withdrawal criteria Any participant can voluntarily withdraw from the study at any time without any compromise to the agreed and proposed treatment. Such a subject will be accounted for during data and statistical analysis. The drop-out sample will not be replaced during the trial. All data pertaining to first time bracket failure will be recorded as agreed until the withdrawal date for an individual sample. The follow up of such a patient will be for orthodontic treatment only and data pertaining to the trial will not be recorded after a sample confirms a withdrawal.
9. Trial termination - reasons for abandoning the trial The trial will be terminated if more than 50% of the brackets fail ( greater than 8 brackets per patient) in the experimental group in at least three patients within the first review appointment (6 weeks). This is because such a high failure rate is clinically unacceptable for continuation of routine orthodontic treatment in the experimental group.
10. Bracket Bonding procedure As the bracket failure rate for the control group has been calculated from a previous study by Littlewood et al., a similar procedure to bond brackets will be followed in this study to avoid intervention bias. All teeth will be bonded including molar teeth. A pre-calibrated light curing unit will be used for setting the glue hard as follows -

CONTROL GROUP

1. 30 second wash and 30 second dry using 3 in 1 syringe
2. 30 second treatment with 37% phosphoric acid gel
3. 30 second wash and 30 second dry using 3 in 1 syringe
4. Application of primer to acid treated enamel and air thinned.
5. Metal bracket placed at long axis point on the outer surface of the tooth
6. Light polymerisation; 30 seconds each on either side of each tooth

   TEST GROUP

<!-- -->

1. 30 second wash and 30 second dry using 3 in 1 syringe
2. 30 second treatment with 37% phosphoric acid gel
3. 30 second wash and 30 second dry using 3 in 1 syringe
4. Metal bracket placed at long axis point on the outer surface of the tooth
5. Light polymerisation; 30 seconds each on either side of each tooth

11. Type of data collected

The following data will be collected:

1. Bracket lost for the first time and subsequent failure with the respective tooth notation
2. Date of bracket failure*
3. Tooth number
4. Whether a primer was used or not
5. Operator involved
6. Time taken from the first step of bonding procedure until the last bracket is placed in each arch
7. Adhesive Remnant Index of debonding interface
8. Patient identification number
9. Length of treatment
10. Peer Assessment Rating score (PAR)

    *If a patient attends an appointment with a bracket failure but the actual failure date cannot be accurately recalled by the patient, then the date of first attendance with bracket failure will be noted.

    12. Outcomes (primary and secondary)

<!-- -->

1. Primary outcome - Bracket failure rate for test and control group
2. Secondary outcomes - Bonding time per bracket, Type of bond failure (using Adhesive Remnant Index), length of treatment and PAR scores.

   Summary of main issues -

   1. PURPOSE AND DESIGN

   Routinely orthodontic treatment is carried out by placing orthodontic brackets on teeth and wires which run through them which help move teeth. These metal brackets are bonded or glued onto the tooth surface by a three step process. Firstly, a mild acid is used to roughen the tooth surface, secondly a free flowing glue (composite primer) is used to fill in the roughened pores and thirdly, the bracket is glued on to the tooth surface with a 'composite' material which sets hard by exposure to a high intensity light. In routine studies, the success of this procedure is measured by bracket failure rates.

   The literature review revealed 7 studies which were relevant to bonding of orthodontic brackets with and without use of primers. Out of these 5 were invitro experimental studies, 1 was a retrospective study and 1 was a prospective non-randomised controlled study. Most studies in this field have been lab based studies which have measured bond strength and failure rates in extracted human teeth. The methodologies used have been retrospective and lack robust study design to eliminate bias. This literature review suggests that the scientific evidence is not clear to indicate whether the use of a primer is absolutely essential to achieve acceptable bracket success/failure rates in a clinical environment. A RCT was designed and carried out in Bradford/Leeds (see previous reference number) which showed no statistical difference between the primer and non primer groups. However, this was a single operator study who was an orthodontic trainee. This study aims for a 'real world' effect by using multiple operators with various degrees of orthodontic experience.

   To summarise, arguably the evidence available from previous studies to either support or refute the use of primer prior to bonding brackets in a clinical setting appears to be weak. The main drawbacks of these studies were related to inconsistent study designs and many of the conclusions may not be applicable for the following reasons -invitro studies, use of chemically cured resins rather than light cured systems which are currently used, different bracket systems, variation in bonding steps, use of flowable composites which are not routinely used for bonding and lack of a prospective randomized controlled study in a clinical setting. All these studies have concluded the need for further research to investigate if clinically acceptable bond strength can be achieved without the use of a primer. If this hypothesis is true, then bonding brackets may become faster, efficient and cost effective. Therefore, a well designed randomized controlled study could be justified to clarify if the use of a primer is essential prior to bonding brackets.

   The results from this randomised clinical trial will help improve our knowledge of the best approach to bonding metal brackets on teeth. If the bracket failure rate is similar in both groups, this suggests that the use of a primer is not always necessary to gain sufficient bond strength in a clinical environment. From a patient's perspective, this would mean lesser clinical time required to place brackets at start of orthodontic treatment. For clinicians and NHS purchasers the outcome of the study will influence clinical chair side time, cost effectiveness (as the primer is the most expensive component in the bonding process) and provide a framework for future studies in this field.

   The trainee student will benefit from training in broad research methodology, scientific critique, statistical concepts and experience in undertaking a randomised clinical trial as a part of Masters project.

   PROTOCOL/ QUALITY ASSURANCE The research will be undertaken as a part of routine orthodontic care provided by a consultant led service in orthodontic departments in Leeds Dental Hospital, St Lukes Hospital and Seacroft hospital. All the patients recruited into the project will receive the same standard of quality orthodontic treatment as provided if they did not choose to partake in the study. All the procedures for orthodontic treatment at the Leeds Dental Institute/Bradford teaching hospitals are quality assured by the Deanery/General Dental Council and Specialist Advisory Committee (SAC) as part of an established three year training programme in Orthodontics (this relates to the fact that one of the researchers will be an orthodontic registrar on on a training pathway). The other clinicians are orthodontic consultants and orthodontic therapists supervised by orthodontic therapists.

   The research committee at Leeds Dental Institute consists of Clinical/Academic Orthodontic Consultants from the region and are routinely involved in supervision of MSc/DDS students regarding their research projects every year. This panel was asked to review the protocol prior to submission and the members include independent reviewers not involved in the study.

   RECRUITMENT All consecutive patients who need fixed appliance therapy will be taken off the NHS waiting list and no attempt will be made to match them for age, sex or malocclusion to ensure a representative sample, except for the exclusion criteria. After informed consent is obtained, they will be randomly allocated to either the control (with Transbond primer) or experimental (without primer) group. This will be done by pre paring opaque numbered sealed envelopes in blocks of 10 in advance by the supervisor (NH) using random number tables. The supervisor will enroll the participants and assign them to their group using the sealed envelopes which blinds the two operators and participants to the assignment before enrollment. Once the envelopes are opened the blinding of the operators will be lost. The operators cannot be blinded in this trial as the intervention administered to the test group cannot be blinded. Treatment will be started on all patients within 3 months of the enrollment.

   INCLUSION / EXCLUSION Inclusion criteria •Patients requiring single or two arch fixed appliance therapy (with no history of previous orthodontic treatment)including patients requiring orthognathic surgery

   •Willing to consent to participate in the trial

   Exclusion criteria
   * Patients with craniofacial anomalies
   * Patients with several buccal restorations or congenital enamel defects
   * Hypodontia cases (with more than one tooth missing in each quadrant)

   CONSENT Children under 16 Routine orthodontic treatment is undertaken at about 12 years of age onwards and a majority of patients requiring orthodontic treatment will be from this age group on a NHS waiting list. These patients have to be included in the study as any clinical relevance of the study will be applicable to patients in this age group, in addition to adults. Appropriate informed consent with parental involvement is routinely followed at the start of treatment for these patients as per NHS trust policy.

   Each participant will be given a patient information sheet outlining the objective, details of the study and answer any frequently asked questions. The patient information sheet will be drafted individually for both adults and children below 16 years of age.

   The informed consent process will be done by the registrar treating the case or the supervising consultant, usually at the next appointment so that enough time is given to the patient if they choose to participate. All participants will be explained regarding the research prior to consent. For participants below 16 years of age, the informed consent process will involve the responsible parent who will sign the form in addition to the child.

   A minimum of 24 hours upto 6 weeks (until the next appointment) of time will usually be available for the patient to think over the decision to participate. In routine orthodontic treatment, usually the registrar/clinician will take treatment records at the initial visit and give a patient information leaflet. Routinely any treatment planning and consent is done at the subsequent appointment which is usually in a few weeks under consultant supervision.

   Any participant requiring language interpretation will be provided with a suitably qualified interpreter, as per the NHS trust protocol. No participant will be excluded on the basis of ethnic origin, language preferences, religion, sexual preference or gender.

   Any involvement of patients with significant learning disability or special needs raises sensitive issues related to comprehension and consent. Although they will be not excluded from participation if they wish to do so, these patients will be offered to partake and the views of the person with parental authority will be considered.

   RISKS, BURDEN AND BENEFITS Possibly, greater failure of brackets (fixed brace attachments) in the experimental group which may need to be glued back on soon after. These failures will not affect the treatment outcome in any way.

   Possibly, extra visit to the department if brackets fail, so that they can be glued back on. This may add on a few weeks of additional time to overall treatment, but will not affect the treatment outcome in any way.

   As per the drafted protocol for the trial " the trial will be terminated if more than 50 % of the brackets fail in the experimental group in at least three patients within the first review appointment (6 weeks). This is because such a high failure rate is clinically unacceptable for continuation of routine orthodontic treatment in the experimental group " In such a situation all the participants will be informed in writing regarding trial termination and all steps would be taken to ensure that routine orthodontic treatment is continued as planned. In such cases all the brackets which have been bonded as per the protocol for the experimental group will be replaced to match the control group i.e. routine treatment.

   CONFIDENTIALITY Each patient will have a patient identification number as per trust policy and this will be quoted on all forms relevant to the study. No other identifiable information will be available on the forms. All electronic data pertaining to the study will be stored in computers within the NHS site and these systems are subject to local NHS trust data protection policies and caldicott principles. No external source will have access to this data. The data will be shared only within the members of the research team for analysis purposes.

   The data will be stored in NHS computers and will be protected as per the NHS trust protocol under the Data Protection Act. The Chief investigator and members of the research team will have access to the data

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients who need fixed appliance treatment will be taken off the waiting list and no attempt will be made to match them for age, sex or malocclusion to ensure a representative sample.

Inclusion criteria is as follows -

* Patients requiring single or two arch fixed appliance therapy (with no history of previous orthodontic treatment)including patients requiring orthognathic surgery
* Willing to consent to participate in the trial

Exclusion Criteria:

* Patients with craniofacial anomalies
* Patients with several buccal restorations or congenital enamel defects
* Hypodontia cases (with more than one tooth missing in each quadrant)

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 156 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Rate of loss of orthodontic brackets | 12 months
  The primary aim of this randomised clinical trial is to investigate if the rate of loss of orthodontic brackets is clinically acceptable when they are bonded onto the tooth surface without the use of a primer as compared to brackets bonded with a conventional primer in adolescent and adult orthodontic patients over a 12 month study period. This will be carried out by multiple operators to ensure a 'real world' orthodontic scenario.

SECONDARY OUTCOMES:
Bonding time per bracket | 12 months
  Bonding time per bracket - This outcome will measure any difference in the time required to bond a single bracket when a primer is not used to a bracket bonded with the conventional three step procedure
Type of failure using adhesive remnant index | 12 months
  Type of bond failure using Adhesive Remnant Index (ARI) - This outcome will measure the type of failure at the bracket-tooth interface, when a bracket fails in either group. The Adhesive Remnant Index is a standardised index which measures the amount of glue which remains over the tooth surface when a bracket fails and thereby categorises the weakest bond area between the tooth-bracket interface.
Length of treatment | 12 months
Peer Assessment rating | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine J Storey, Principal Investigator — University of Leeds; Simon J Littlewood, Study Director — University of Leeds; Nadine Houghton, Study Director — University of Leeds